CLINICAL TRIAL: NCT01799226
Title: Study of the Anti-Inflammatory Effects of Colgate Total® During an Experimental Gingivitis Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Janet Kinney, Assistant Professor of Dentistry, Director of Dental Hygiene Program, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HUM00055445
Record Dates: First submitted 2013-02-24; First posted 2013-02-26 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Toothpastes; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toothpaste without Triclosan (Active Comparator): This arm will use a toothpaste that does not contain triclosan
  Interventions: Other: Toothpaste without triclosan
- Triclosan (Experimental): This arm will use colgate total which contains triclosan
  Interventions: Other: Triclosan

INTERVENTIONS:
Other: Toothpaste without triclosan — this intervention will use a toothpaste without triclosan
  Arms: Toothpaste without Triclosan
Other: Triclosan — this intervention will use Colgate Total which contains triclosan
  Other Names: Colgate total toothpaste
  Arms: Triclosan

SUMMARY:
This study evaluates the anti-inflammatory effects of Colgate Total® during an experimental gingivitis model developed by Löe et al. Half of the participants will use Colgate Total® (which contains triclosan), while the other half will use a toothpaste which does not contain triclosan as the control.

DETAILED DESCRIPTION:
This will be a double-blind. Subjects will be randomly assigned to the test or control dentifrice arm. Enrolled subjects will also be randomly assigned to either right or left side mandibular stent.

During the induction phase (i.e., day 0 to day 21), participants are instructed to refrain from all hygiene procedures in the stent area. During this time period, participants evenly distributed 2mL of their assigned dentifrice into their stent, allowing it to come into contact with the areas of experimental gingivitis for two minutes twice daily while traditional tooth brushing was performed in the non-stent areas. Clinical measures, saliva, gingival crevicular fluid and plaque samples will be collected at days 0, 14, 21, and 35 study visits. A randomization chart will be used to identify which two sites (teeth and tooth surface) will be used at the specific study visit for collection of gingival crevicular fluid(GCF) and plaque.

ELIGIBILITY:
Inclusion Criteria:

* Race - all
* Gender - female or male
* Age - 18 to 40 years old
* Dentition - minimum of 20 permanent teeth
* Probing Pocket Depth of 1-4mm in all sites
* Mean Clinical Attachment Levels of 2mm on all teeth
* Bleeding Upon Probing of greater than 30% at Day -14 Study Visit
* Consent Form - read, understood, and signed
* Study Procedures - willing to follow all study procedures
* At Day 0 Study Visit, all subjects must have a BOP of less than 10%. Subjects not meeting the BOP study criteria will be asked to return in 2 weeks for a second assessment visit. Subjects who do not meet the inclusion criteria
* BOP less than 10% at the second assessment visit will be exited from the
* study

Exclusion Criteria:

* Medical History - a history of alcoholism or drug abuse
* Diseases of the immune system
* Medical condition that may affect outcome (neurologic or psychiatric disorders, systemic infection
* Medications - chronic medications known to affect the periodontal status (calcium antagonists anticonvulsives, immunosuppressives, anti-inflammatory medications, phenytoin, Depo-Provera contraceptive injection users
* New oral contraceptives users within 3 months of baseline or are planning on starting oral contraceptives during the study
* Hypersensitivity - previous known reaction to or oral allergy to any ingredient in the study toothpaste
* Antibiotics - antibiotic therapy within 3 months of baseline visit
* antibiotic therapy needed for infective endocarditis prophylaxis or total joint replacement
* Use of antiseptics - homecare regime using products to control dental plaque formation within 30 days prior to baseline visit
* Smoking - current smokers, smokers who quit smoking less than one year ago, or a pack-year history of more than or equal to 10 (pack-years will be calculated by multiplying the number of years smoked by the average number of cigarette packs smoked per day)
* Continine - positive urine analysis results
* Current Dental Treatment - orthodontic or periodontal treatment
* Untreated Dental Treatment - untreated carious lesions
* Defective restorations which could exacerbate during a period of oral hygiene abstinence
* Pregnant or women breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kinney, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Pancer BA, Kott D, Sugai JV, Panagakos FS, Braun TM, Teles RP, Giannobile WV, Kinney JS. Effects of triclosan on host response and microbial biomarkers during experimental gingivitis. J Clin Periodontol. 2016 May;43(5):435-44. doi: 10.1111/jcpe.12519. Epub 2016 Apr 6. PMID 26820239

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially 15 participants were sought for each arm, but when two were withdrawn from the control arm, two more participants were recruited and randomized, one to each arm. So total start on each arm was 16.
  The Disqualification noted below for one participant was because s/he no longer met inclusion criteria as of day 14.
Groups:
- Control Arm: Participants were randomly assigned to either the test (triclosan dentifrice) or control (fluoride dentifrice) arm of the study and to either the right or left stent side. The control dentifrice was composed of 0.76% sodium monofluorophosphate 1000 ppm (0.15% w/v fluoride ion) as the active ingredient along with inactive ingredients (Colgate® Cavity Protection Great Regular Flavor Fluoride Toothpaste).
- Test Arm: Participants were randomly assigned to either the test (triclosan dentifrice) or control (fluoride dentifrice) arm of the study and to either the right or left stent side. The test dentifrice was composed of 0.24% sodium fluoride 1100 ppm 0.243% (0.14% w/v fluoride ion) and triclosan 0.30% in combination with 2% polyvinyl methyl ether maleic acid copolymer as the active ingredients along with inactive ingredients (Colgate® Total® Clean Mint Paste).
Period: Overall Study
Arm/Group | Control Arm | Test Arm
Started | 16 | 16
Right Stent Side | 8 | 8
Left Stent Side | 8 | 8
Completed | 14 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disqualified at Day 14 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data analysis only included examining the test (triclosan dentifrice) or control (fluoride dentifrice).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Test Arm | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Customized [Mean (Full Range); unit: years]
  Age | 27.07 [21.92 to 32.32] | 26.06 [20.83 to 31.29] | 26.57 [20.83 to 32.32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 2 | 7 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Bleeding on probing ≤ 10% [Mean (Full Range); unit: Percent of sites bleeding on probing] | 0.065 [0.02 to 0.10] | 0.063 [0.02 to 0.10] | 0.064 [0.02 to 0.10]

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Gingival Index (Loe & Silness 1963) to Day 35
Description: Loe & Silness 1963 is a score of 0-3 with 0 = Absence of inflammation, 1 = Mild inflammation, slight change in color and texture, 2 = Moderate inflammation, glazing, redness, edema and hypertrophy, 3 = Severe inflammation, redness and hypertrophy, ulceration. This index was used at days 0, 14, 21 and 35.
Time Frame: Baseline to 35 Days
Population: Data analysis only included examining the test (triclosan dentifrice) or control (fluoride dentifrice).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Arm | Test Arm
Number analyzed (Participants) | 14 | 16
units on a scale
  Gingival index Baseline | 0.25 (0.04) | 0.32 (0.03)
  Gingival index Day 14 | 1.33 (0.06) | 1.38 (0.07)
  Gingival index Day 21 | 1.56 (0.07) | 1.52 (0.07)
  Gingival index Day 35 | 0.39 (0.07) | 0.47 (0.07)

2. Primary Outcome: Change From Baseline in Plaque Index (Silness & Loe 1964) to Day 35
Description: Silness & Loe 1964 is a score of 0-3 with 0 = No plaque, 1 = A film of plaque adhering to free gingival margin and adjacent area of tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface, 2 = Moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin, which can be seen with the naked eye, 3 = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin. This index was used at days 0, 14, 21 and 35.
Time Frame: Baseline to 35 Days
Population: Data analysis only included examining the test (triclosan dentifrice) or control (fluoride dentifrice).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Arm | Test Arm
Number analyzed (Participants) | 14 | 16
units on a scale
  Plaque index Baseline | 0.37 (0.06) | 0.44 (0.07)
  Plaque index Day 14 | 1.24 (0.07) | 1.49 (0.08)
  Plaque index Day 21 | 1.84 (0.10) | 1.81 (0.10)
  Plaque index Day 35 | 0.45 (0.06) | 0.57 (0.04)

3. Other Pre Specified Outcome: Unstimulated Whole Saliva Will be Collected for Inflammatory Biomarker Expression.
Description: Inflammatory biomarker expression will be quantified using a custom human 10-complex protein array that is optimized for sensitivity, specificity, stability, and intraassay coefficient of variation by comparing to single cytokine enzyme-linked immunosorbent assays (Quantibody Custom Array, RayBiotech, Norcross, GA).
Time Frame: Baseline to 35 Days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Plaque Samples Will be Collected for Bacterial Species Detection.
Description: Supra- and sub-gingival plaque samples will be gently collected using a sterile curet and a one stroke method from two randomized sites within the stent area. The detection of 40 bacterial species will be evaluated by the checkerboard DNA-DNA hybridization technique originally described by Socransky et al. 1994.
Time Frame: Baseline to 35 Days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Gingival Crevicular Fluid (GCF) Will be Collected for Inflammatory Biomarker Expression.
Description: A total of 10 biomarkers will be analyzed based on the results from Lee and colleagues: IL-1α, IL-1β, IL-6, IL-8, IL-10, MCP-1, MMP-8, MMP-9, TIMP-1, and TIMP-2.
Time Frame: Baseline to 35 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse event data was collected for 9 months.
Description: Data analysis only included examining the test (triclosan dentifrice) or control (fluoride dentifrice).
Arm/Group | Control Arm | Test Arm
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=16) | Test Arm (N=16)
Aphthous ulcer (General disorders) | 1 (1) | 3 (3)
Tissue slough (General disorders) | 2 (2) | 0 (0)
TMJ soreness (General disorders) | 0 (0) | 1 (1)
Tooth decay (General disorders) | 1 (1) | 0 (0)
Tingling in tongue (General disorders) | 0 (0) | 1 (1)
Toothbrush trauma (General disorders) | 0 (0) | 1 (1)
Herpetic lesion (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No